CLINICAL TRIAL: NCT05574218
Title: Effect of a Maintenance Protocol Based on the Surgical Treatment of Peri-implantitis and Implant Surface Decontamination With Glycine Powder Air-polishing
Brief Title: Effect of a Maintenance Protocol After Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS/MTO
Record Dates: First submitted 2022-09-26; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Investigator

ARMS (2):
- Glycine - Test (Experimental): Polishing treatment with glycine powder air-polishing after ultrasonic plaque debridement.
  Interventions: Procedure: Glycine air powder
- Rubber cup - Control (Active Comparator): Polishing treatment with a rubber cup and polishing paste after ultrasonic debridement
  Interventions: Procedure: Rubber cup polishing

INTERVENTIONS:
Procedure: Glycine air powder — Every 3 months, ultrasonic instrumentation was carried out with an specific implant tip coated with Polyether Ether Ketone (PEEK), activated subgingivally and circumferentially around the implant. Then, the implants were treated with glycine powder air-polishing.
  Arms: Glycine - Test
Procedure: Rubber cup polishing — Every 3 months, ultrasonic instrumentation was carried out with an specific implant tip coated with Polyether Ether Ketone (PEEK), activated subgingivally and circumferentially around the implant. Then, the implants were treated with rubber cup and a polishing paste.
  Arms: Rubber cup - Control

SUMMARY:
This study was designed as a 12-month, two arms, randomized clinical trial to evaluate the efficacy of a supportive treatment protocol (SPIT). Thirty patients were randomized, six months after access-flap surgery, in two different SPIT groups. After ultrasonic debridement, the affected implant surfaces of the test group were treated with glycine powder air-polishing, while implants in the control group a rubber cup and polishing paste was used. Maintenance visits were carried every 3 months and clinical, radiological, microbiological and biochemical variables were registered at baseline (6 months after surgery) and after a follow-up period of 12 months (18 months after surgery).

DETAILED DESCRIPTION:
Study design:

This study was designed as a 12-month, two arms, RCT to evaluate the efficacy of a SPIC protocol. Thirty patients were randomized, six months after access-flap surgery, in two different SPIT groups. After ultrasonic debridement, the affected implant surfaces of the test group were treated with glycine powder air-polishing, while implants in the control group a rubber cup and polishing paste was used. Maintenance visits were carried every 3 months and clinical, radiological, microbiological and biochemical variables were registered at baseline (6 months after surgery) and after a follow-up period of 12 months (18 months after surgery).

Interventions:

At the 6-month evaluation after the surgery, the baseline data for the present study were obtained and patients were randomised using a computerized block randomization protocol to one of the following SPIC protocols. In the test group, implant surfaces were treated with glycine powder air-polishing after ultrasonic instrumentation; the specific nozzle was activated subgingivally and circumferentially around the implant for 1 minute. In the control group, implants were cleaned with a rubber cup and polishing paste after ultrasonic instrumentation. This SPIC visits were carried out at 6 (baseline visit), 9, 12, 15 and 18 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one implant with peri-implantitis, defined as: radiographic evidence of bone loss >2 mm, inflammation of the peri-implant mucosa as defined by positive BoP and/or suppuration, and at least one site with PD ≥ 5 mm.
* Based on the radiographic examination, the affected implant should not have a vertical peri-implant defect. Positive selection was based on the presence of pe-ri-implant lesions wider than 4 mm, with an angle greater than 35 º.
* In patients with a history of periodontitis, periodontal therapy should have been provided at least 6 months prior to the initiation of the study.

Exclusion Criteria:

* Presence of relevant medical conditions and/or systemic medications that would contraindicate the surgical procedure or modify the tissue response after therapy.
* Patients requiring antibiotic prophylaxis.
* Heavy smokers (> 10 cigarettes/day).
* Pregnant or lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | Baseline, 6 and 18 months after the surgical procedure
  Changes in Probing Pocket Depth measured in milimeters with a manual periodontal probe

SECONDARY OUTCOMES:
Distance of Gingival Recession | Baseline, 6 and 18 months after the surgical procedure
  Recession distance of the mucosal margin relative to the restoration margin (REC) at the implant (6 sites/implant) measured in milimeters with a manual periodontal probe
Bleeding on Probing index | Baseline, 6 and 18 months after the surgical procedure
  Rate of Presence / absence Bleeding on Probing at the implant (6 sites/implant)
Plaque Index | Baseline, 6 and 18 months after the surgical procedure
  Rate of Presence / absence of Plaque at the implant (6 sites/implant)
Suppuration Index | Baseline, 6 and 18 months after the surgical procedure
  Rate of Presence / absence of suppuration at the implant (6 sites/implant)
Radiographic bone loss distance measured from the prosthetic connection platform to the bottom of the intraosseous defect | Baseline, 6 and 18 months after the surgical procedure
  Intraoral standardised radiographs of the site of interest measured in digital intraoral radiographs using an image-processing software
Concentration of the selected cytokines measured in pg/ml (IL1B; Il-6; IL-8; Tumoral Necrosis Factor Alpha) | Baseline, 6 and 18 months after the surgical procedure
  Samples taken from the gingival crevicular fluid (GCF) were taken from each included implant from the deepest PD site with positive BoP, at baseline and at the final evaluation, always prior to microbiological sampling. Samples were taken using the filter paper technique. After isolation of the area with cotton rolls and gentle cleaning with air and a gauze to remove supragingival biofilm deposits and potential saliva contamination, a paper strip of standard length and height was inserted into the peri-implant pocket, until mild resistance was felt and left in place for 30 seconds. The soaked volume of GCF was measured using the Periotron 8000® device. Subsequently, the paper strips were inserted in micro-centrifuge plastic tubes and immediately stored at -80°C until further processing. Analyses were carried out using a Luminex System (Luminex® 200, Luminex Corporation, Austin, TX, USA) to determine volume of the following biomarkers: IL-1β, IL-6, IL-8 and TNF-α.
Presence of putative periodontal pathogens | Baseline, 6 and 18 months after the surgical procedure
  Sample from the deepest site in the evaluated implant using two consecutive sterile paper-points kept in place for 10 seconds and then transferred into a screw-capped vial, containing 1.5 mL of reduced transport fluid (RTF). Samples were transferred to the microbiological laboratory within 2 hours and homogenized by vortexing for 30 seconds and serially diluted in phosphate buffer saline (PBS). Then, 0.1 mL of each dilution was plated manually on the specific medium Dentaid-1, for the detection of Aggregatibacter actinomycetemcomitans, and incubated for 3 days in air with 5% CO2 at 37ºC. Samples were also plated into a non-selective blood agar plate, supplemented with haemine (5 mg/l), menadione (1 mg/l) and 5% sterile horse blood, with 7-14 days of anaerobic incubation.
Frequency of detection of putative periodontal pathogens | Baseline, 6 and 18 months after the surgical procedure
  Sample from the deepest site in the evaluated implant using two consecutive sterile paper-points kept in place for 10 seconds and then transferred into a screw-capped vial, containing 1.5 mL of reduced transport fluid (RTF). Samples were transferred to the microbiological laboratory within 2 hours and homogenized by vortexing for 30 seconds and serially diluted in phosphate buffer saline (PBS). Then, 0.1 mL of each dilution was plated manually on the specific medium Dentaid-1, for the detection of Aggregatibacter actinomycetemcomitans, and incubated for 3 days in air with 5% CO2 at 37ºC. Samples were also plated into a non-selective blood agar plate, supplemented with haemine (5 mg/l), menadione (1 mg/l) and 5% sterile horse blood, with 7-14 days of anaerobic incubation.
Proportions of putative periodontal pathogens | Baseline, 6 and 18 months after the surgical procedure
  Sample from the deepest site in the evaluated implant using two consecutive sterile paper-points kept in place for 10 seconds and then transferred into a screw-capped vial, containing 1.5 mL of reduced transport fluid (RTF). Samples were transferred to the microbiological laboratory within 2 hours and homogenized by vortexing for 30 seconds and serially diluted in phosphate buffer saline (PBS). Then, 0.1 mL of each dilution was plated manually on the specific medium Dentaid-1, for the detection of Aggregatibacter actinomycetemcomitans, and incubated for 3 days in air with 5% CO2 at 37ºC. Samples were also plated into a non-selective blood agar plate, supplemented with haemine (5 mg/l), menadione (1 mg/l) and 5% sterile horse blood, with 7-14 days of anaerobic incubation.
Counts of putative periodontal pathogens | Baseline, 6 and 18 months after the surgical procedure
  Sample from the deepest site in the evaluated implant using two consecutive sterile paper-points kept in place for 10 seconds and then transferred into a screw-capped vial, containing 1.5 mL of reduced transport fluid (RTF). Samples were transferred to the microbiological laboratory within 2 hours and homogenized by vortexing for 30 seconds and serially diluted in phosphate buffer saline (PBS). Then, 0.1 mL of each dilution was plated manually on the specific medium Dentaid-1, for the detection of Aggregatibacter actinomycetemcomitans, and incubated for 3 days in air with 5% CO2 at 37ºC. Samples were also plated into a non-selective blood agar plate, supplemented with haemine (5 mg/l), menadione (1 mg/l) and 5% sterile horse blood, with 7-14 days of anaerobic incubation.

IPD SHARING:
Plan to Share IPD: No